CLINICAL TRIAL: NCT06960005
Title: Screening and Exercise Intervention to Improve Muscle Performance, Reduce Risk of Falls, and Enhance Quality of Life in Thyroid Hormone Disease: ThyMoves
Brief Title: ThyMoves: Screening and Exercise to Improve Muscle, Enhance Quality of Life, and Reduce Fall Risk in Thyroid Disease
Acronym: ThyMoves
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Steno Diabetes Center Nordjylland (Other)
Responsible Party: Principal Investigator, Mia Daugaard Madsen, Principal Investigator, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20240055
Record Dates: First submitted 2025-04-02; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Disease; Hashimoto's Thyroiditis; Hyperthyreosis and Goiter; Hypothyroidism
Keywords: Health-related Quality of Life; Exercise intervention
MeSH Terms: conditions — Thyroid Diseases; Goiter; Hypothyroidism | interventions — Activities of Daily Living

STUDY DESIGN:
Intervention Model Description: Screening and exercise intervention with Rhythm- and Multitask-Based Activity (RYMA) and Activities of Daily Living (ADL)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise intervention: RYMA (Experimental): Participants in this arm will engage in the Rhythm- and Multitask-Based Activity (RYMA) program, a 26-week multicomponent exercise intervention designed to enhance quality of life, improve physical function, and prevent falls. The program integrates strength, balance, coordination, and cognitive-motor training, along with Activities of Daily Living (ADL)-based exercises to support real-world functionality.
  Interventions: Other: Rhythm- and Multitask-Based Activity (RYMA) and Activities of Daily Living (ADL)
- Control group: Usual Care/No Structured Exercise Intervention (No Intervention): Participants will be screened and followed but not participate in the exercise intervention and continue their usual activities.

INTERVENTIONS:
Other: Rhythm- and Multitask-Based Activity (RYMA) and Activities of Daily Living (ADL) — Participants will engage in one-hour exercise sessions twice weekly for 26 weeks: one day of RYMA training and one day of ADL-based training
  Arms: Exercise intervention: RYMA

SUMMARY:
Objectives:

This study aims to assess health-related quality of life (QoL) in adults with thyroid hormone disorders and identify modifiable factors to improve QoL in patients with Hashimoto's thyroiditis (HT) and multinodular toxic goiter (MNTG) through an exercise intervention.

Primary Outcome:

1. Assess the impact of a tailored exercise program on health-related QoL in patients with HT and MNTG using the ThyPRO questionnaire.

Secondary Outcomes:

1. Evaluate the need for a screening tool to identify thyroid patients with reduced health-related QoL despite being euthyroid.
2. Assess the impact of the exercise intervention on body composition, strength, and balance function in HT and MNTG patients.

Methods:

The study is a combined cross-sectional survey and randomized controlled trial into the health related QoL in patients diagnosed with thyroid hormone disease. The cross-sectional survey will assess the overall health-related QoL in patients diagnosed with thyroid hormone disease, and help identify eligible participants for the subsequent RCT.

The RCT will evaluate the efficacy of a comprehensive screening and exercise intervention in patients ≥ 65 years diagnosed with HT or MNTG, experiencing reduced health-related QoL.

Participants:

The aim is to recruit 74 patients with HT and 74 patients with MNTG, including 50 participants from each group with reduced health-related QoL (defined in this study as ThyPRO score ≥ 30) and 24 with good health-related QoL (ThyPRO score ≤ 20)

ELIGIBILITY:
Inclusion Criteria:

1. Women with minimum 65 years of age, with no upper limit.
2. Verified diagnosis of HT or MNTG
3. Euthyroid for at least 6 months
4. Signed the informed consent

Exclusion Criteria:

1. Current participation in a structured exercise program or regular physical exercise activity above 5 hours per week
2. Previous experience with rhythm-based multitask exercise.
3. Diagnosed with significant neurological diseases (e.g. Multiple Sclerosis and myasthenia gravis), vestibular diseases or newly orthopedic surgeries (e.g. knee or hip replacement)
4. Fully dependent on walking aids
5. Active malignancy or terminal illness
6. Inability to understand Danish written and/or verbally
7. Having severely impaired cognitive function, defined as a score below 8 on the cognitive assessment "the short orientation-memory-concentration test"
8. Treatment with amiodarone within the last year
9. No changes within the last six months in medications affecting weight or body composition - e.g., GLP-1 electrolyte/fluid balance - e.g., diuretics or corticosteroid
10. Participation in other clinical intervention studies within the last six months

For the cross sectional survey:

Inclusion criteria:

1. Men and women with a minimum of 18 years
2. Diagnosis of primary hypothyroidism or primary hyperthyroidism

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 148 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life after the Exercise Intervention | 26 weeks and 52 weeks
  The Thyroid-Related Quality of Life Measure questionnaire (ThyPRO) consists of 85 items summarized into 13 scales and one single item measuring the overall impact of thyroid disease on quality of life. It includes questions on symptoms, mood, memory, tiredness, and general health. Each item is rated on a 0-4 Likert scale, with scores transformed to a 0-100 scale; higher scores indicate worse health status.
  The ThyPRO questionnaire wil be used to assess changes in health-related QoL at 26 weeks (post-intervention) and 52 weeks (follow-up).

SECONDARY OUTCOMES:
Changes in Muscle Mass | 26 weeks and 52 weeks
  Full body Dual-Energy X-ray Absorptiometry (DXA) scans will be used to assess changes in muscle mass. These outcomes will evaluate whether the intervention influences muscle quality over time, with comparisons between intervention and control groups
Changes in Fat Mass Distribution | 26 weeks and 52 weeks
  Full-body DXA scans will be used to assess changes in fat mass distribution over time. Comparisons will be made between intervention and control groups
Muscle Strength | 26 weeks and 52 weeks
  Change in muscle strength assessed by handgrip strength and isometric knee extension strength (using a dynamometer).
Balance Function | 26 weeks and 52 weeks
  Change in balance function assessed through Center of Pressure (CoP).
Identification of Patients with Reduced Health-Related Quality of Life | Baseline (Day 1)
  To assess the potential need for future implementation of health-related quality of life (HRQoL) screening in patients with thyroid hormone disease, based on the number of patients identified with reduced HRQoL using the Thyroid-Related Quality of Life Questionnaire (ThyPRO). The ThyPRO includes 85 items across 13 scales and one overall impact item. Scores range from 0 to 100, with higher scores indicating worse health status.

OTHER OUTCOMES:
Improvement in Nerve Function | Baseline, 26 weeks and 52 weeks
  To estimate the change in nerve fiber function by assessing small, large, and autonomic neuropathy using standardized neurophysiological methods following the exercise intervention in patients with HT and MNTG.
Reduction in fall rates | 26 weeks and 52 weeks
  To estimate changes in fall rates in patients aged >65 with HT or MNTG following the RYMA intervention, compared to their baseline measures (self-controls) and to a usual care group (no RYMA).

CONTACTS AND LOCATIONS:
Locations (1):
- Diabeteshuset, Gistrup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided